CLINICAL TRIAL: NCT03055507
Title: Effect of Post-operative Ibuprofen After Surgery for Chronic Rhinosinusitis: A Prospective, Pilot, Cohort Study
Brief Title: Effect of Post-operative Ibuprofen After Surgery for Chronic Rhinosinusitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Craig Miller, Resident, School of Medicine: Otolaryngology-Head & Neck Surgery, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000798
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Ibuprofen; Acetaminophen; Oxycodone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard pain regimen of acetaminophen 650 mg q6hrs while awake until cessation of need for scheduled pain medication with the addition of oxycodone 5 mg q3 hrs PRN (as needed) pain.
  Interventions: Drug: Acetaminophen 650 mg; Drug: OxyCODONE 5 Mg Oral Tablet
- Ibuprofen (Experimental): Alternating every 3 hours acetaminophen 650 mg and ibuprofen 400 mg while awake until cessation of need for schedule pain medication with the addition of oxycodone 5 mg q3hr PRN pain.
  Interventions: Drug: Ibuprofen 400 mg; Drug: Acetaminophen 650 mg; Drug: OxyCODONE 5 Mg Oral Tablet

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Addition of ibuprofen to standard pain regimen.
  Other Names: Motrin
  Arms: Ibuprofen
Drug: Acetaminophen 650 mg — Standard analgesic provided post-operatively to patients undergoing sinus surgery
  Other Names: Tylenol; Paracetamol
Drug: OxyCODONE 5 Mg Oral Tablet — Standard PRN medication offered post-operatively for breakthrough pain

SUMMARY:
Endoscopic sinus surgery (ESS) for chronic rhinosinusitis (CRS) is a common procedure in the US, with about 250,000 cases performed annually. Currently, there is no consensus, evidence-based post-operative pain regimen; with the majority of practitioners opting for a combination of acetaminophen and narcotics for pain control. Most rhinologists avoid NSAIDs due to decreased platelet aggregation and the theoretical risk of increased post-operative bleeding. No studies to date have evaluated the use of ibuprofen in CRS patients following ESS. Additionally, there is a lack of information regarding the average narcotic requirement following ESS.

The purpose of this pilot prospective cohort study is to evaluate the use of narcotics in sinus surgery and the effect of ibuprofen in the non-packed nose following ESS. This investigation will help to gain understanding of current opioid use in post-op sinus patients and assess the safety and effectiveness of post-operative ibuprofen administration on pain. The investigators aim to quantify the average narcotic use following ESS, as well as evaluate the effect of the addition of ibuprofen to the standard analgesic regimen on pain scores and post-operative epistaxis. The investigators hypothesize that the use of ibuprofen will decrease pain scores on a 10-cm visual analogue scale when compared with individuals who do not use ibuprofen post-operatively, this will lead to decreased opioid use in the post-operative period. Additionally, the investigators hypothesize no increase in post-operative bleeding rates, again based on a 10-cm visual analogue scale and bleeding events.

In summary, this will be the first study to the investigators knowledge to examine the effect of post-operative ibuprofen use and its effects on opioid use, as well as pain and epistaxis outcomes, in ESS. By performing this pilot prospective cohort study, the investigators will be equipped to design and perform the optimal prospective, randomized study evaluating the effect of NSAID in ESS during the post-operative period. The overarching goal of this investigation is to decrease opioid use in post-operative pain control following ESS.

DETAILED DESCRIPTION:
Opioid use and abuse is a major public health issue. US Surgeon General, Dr. Vikta Murthy, has recently called for investigation into evidence-based prescribing of opioids. Endoscopic sinus surgery (ESS) for chronic rhinosinusitis (CRS) is a common procedure in the US, with about 250,000 cases performed annually.1 Currently, there is no consensus for appropriate post-operative analgesic control after ESS. Many practitioners use a combination of acetaminophen and narcotics for pain control. Importantly, most rhinologists avoid the use of NSAIDs due to a theoretical concern for decreased platelet aggregation and the potential risk of increased post-operative hemorrhage. However, no studies to date have evaluated the use of ibuprofen in CRS patients following ESS. Conceivably, if the investigators can improve post-operative pain control after ESS with using ibuprofen, then that may decrease standard prescriptions for narcotic analgesics. Given that 60% of narcotic overdose deaths are due to prescribed medications, this would help deliver improved pain control with less narcotic prescriptions. Therefore, the objective is to perform a pilot prospective cohort study to evaluate the use of narcotics in sinus surgery and the effect of ibuprofen following ESS. This pilot study will provide critical baseline data for narcotic use, ibuprofen safety and ibuprofen analgesic impact to optimize the design of a future prospective, randomized study. Thus, specific aims are as follows:

Specific Aim 1: Patients with CRS will document their narcotic use in the first 7 days following sinus surgery. This will allow us to reform prescribing practices. Hypothesis: There will be a wide range of narcotic usage among post-op patients with the mean usage being less than the amount typically prescribed post-operatively.

Specific Aim 2: During enrollment the investigators will ask patients to self-select the study arm they would like to join (ibuprofen versus no ibuprofen) thus documenting willingness to participate, which is important in designing the future randomized study. Hypothesis: Most patients approached will be wiling to participate and will indicate willingness to be part of a similar randomized study.

Specific Aim 3a: Determine impact of ibuprofen on post-operative sinus surgery patients' pain level. The investigators will analyze patients with CRS that are set to undergo ESS in two cohorts (standard pain regimen and standard pain regimen plus ibuprofen) and assess postoperative pain at days 1, 3, and 7 by 10-cm visual analogue scale, amount of post-operative narcotic pain medication used, and number of days post-operatively taking narcotic medications, Hypothesis: Addition of ibuprofen will decrease post-operative pain and will decrease number of opioid pills used.

Specific Aim 3b: Determine impact of ibuprofens impact on post-operative epistaxis. Using the same patient cohorts, degree of epistaxis will be assessed utilizing standardized recording documents and a 10-cm visual analogue scale, as well as a previously used epistaxis grading system.2 The investigators will assess these outcomes on post-operative day 1, 3, and 7. Hypothesis: Addition of ibuprofen will demonstrate no increase in post-operative epistaxis compared to the control group.

At the study institution, approximately 250 endoscopic sinus cases are performed per year performed by two rhinologists. This will yield ample potential research subjects to complete the study. To the investigators knowledge, there is one previous study looking at the effect of peri-operative NSAIDs during ESS. This study found no increased risk in intraoperative or postoperative bleeding after administration of ketorolac. This will be the first study to examine the effect of post-operative oral ibuprofen use and its effects on opioid use, as well as pain and epistaxis outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRS scheduled to undergo functional endoscopic sinus surgery
* >18 years old
* Able to speak and comprehend written English

Exclusion Criteria:

* Contraindication to NSAID use (Chronic kidney disease, Peptic Ulcer disease, Aspirin exacerbated respiratory disorder (AERD), etc.)
* Previous history of bleeding disorder
* Sinus cancer
* Cystic Fibrosis
* Current use of anti-coagulant or anti-platelet medication (during and immediately after ESS)
* History of chronic pain, fibromyalgia, or opioid addiction
* Excessive bleeding during the surgery as determined by the attending surgeon
* Contraindication to acetaminophen use
* Daily use of analgesics including ibuprofen, other NSAIDs, acetaminophen, narcotic medications or other analgesics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Miller, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard pain regimen of acetaminophen 650 mg q6hrs while awake until cessation of need for scheduled pain medication with the addition of oxycodone 5 mg q3 hrs PRN pain.
  Acetaminophen 650 mg: Standard analgesic provided post-operatively to patients undergoing sinus surgery
  OxyCODONE 5 Mg Oral Tablet: Standard PRN medication offered post-operatively for breakthrough pain
Period: Overall Study
Arm/Group | Control | Ibuprofen
Started | 16 | 26
Completed | 16 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ibuprofen | Total
Number analyzed (Participants) | 16 | 26 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16) | 53 (18.5) | 49 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 8 | 12 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 26 | 42
Chronic rhinonsinusitis (CRS) with Nasal Polyposis [Count of Participants; unit: Participants] | 1 | 12 | 13
Duration of surgery [Mean (Standard Deviation); unit: minutes] | 90 (44.2) | 91 (49.1) | 90 (46)
Estimated blood loss [Mean (Standard Deviation); unit: milliliters] | 49 (34.7) | 51 (22.6) | 51 (30)
Lund-MacKay CT grading Score [Mean (Standard Deviation); unit: units on a scale] — method for radiologic staging of chronic rhinosinusitis.
  When reading a CT scan of the paranasal sinuses and ostiomeatal complex, the reader assigns each sinus a score of:
  0 (no abnormality)
  1. (partial opacification) or
  2. (complete opacification) The osteomeatal complex (OMC) is assigned a score of either 0 (not obstructed) or 2 (obstructed).
  The sinuses are grouped into:
  frontal sinus anterior ethmoidal cells posterior ethmoidal cells maxillary sinus sphenoid sinus OMC
  Scale ranges from 0-24. Score is sum of each group. Higher values represent more severe disease.
  units on a scale | 9.4 (6) | 10.1 (6) | 9.8 (6)
Sinonasal outcome test-22 score (SNOT-22) [Mean (Standard Deviation); unit: units on a scale] — Baseline test of CRS symptoms. Previously validated widely used scale for CRS symptoms.
  This is a patient reported outcome scale. Each of 22 subdomains scored on a scale of 0-5. 0 indicating no problem, 5 indicating problem as bad as can be.
  Scores range from 0 to 110.
  Higher scores reflect worse symptoms.
  units on a scale | 44 (22.6) | 42 (18.9) | 42 (19.7)
Number of sinuses operated [Mean (Standard Deviation); unit: sinuses] | 5.3 (2.4) | 5.9 (1.8) | 5.7 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analogue Scale (VAS)
Description: 10-cm visual analogue scale used to indicate level of post-operative pain. 0 indicates no pain and 10 indicates worst pain imaginable.
Time Frame: Post-operative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 16 | 26
units on a scale | 3.3 (2.1) | 2.3 (2.1)
Statistical Analysis 1: Comparison: Control vs Ibuprofen; Test type: Superiority; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = -0.9, 96% CI 2-sided [-2.4 to 0.5]

2. Primary Outcome: Pain Visual Analogue Scale
Description: 10-cm visual analogue scale used to indicate level of post-operative pain. 10-cm visual analogue scale used to indicate level of post-operative pain. 0 indicates no pain and 10 indicates worst pain imaginable.
Time Frame: Post-operative day 3
Population: Patients undergoing sinus surgery stratified into study arms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 16 | 26
units on a scale | 3.0 (2.1) | 1.7 (1.4)

3. Primary Outcome: Pain Visual Analogue Scale
Description: 10-cm visual analogue scale used to indicate level of post-operative pain. Scale from 0-10 with 0 indicating no pain and 10 indicating worst pain imaginable.
Time Frame: Post-operative day 7
Population: Same as previous
Measure: Mean (Standard Deviation); unit: units on the pain visual analogue scale
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 16 | 26
units on the pain visual analogue scale | 3.3 (2.1) | 2.3 (2.1)

4. Secondary Outcome: Number of Opioid Pills
Description: Number of opioid pills taken daily following surgery
Time Frame: Post-operative days 1-7
Measure: Mean (Standard Deviation); unit: pills per day
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 16 | 24
pills per day | 4 (1) | 4 (1)

5. Secondary Outcome: Bleeding Visual Analogue Scale
Description: 10-cm visual analogue scale used to indicate amount of nasal bleeding post-operatively. 0 = no bleeding, 10 = life-threatening bleeding
Time Frame: Post-operative days 1, 3, and 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 15 | 24
units on a scale
  Post-operative day 1 | 3.2 (2.0) | 2.3 (2.1)
  Post-operative day 3 | 3.2 (2.1) | 2.3 (1.8)
  Post-operative day 7 | 1.2 (0.6) | 0.5 (1.1)

6. Secondary Outcome: 0-4 Bleeding Scale
Description: Previously used 0-4 scale to indicate amount of nasal bleeding. 0 indicating no bleeding and 4 indicating life threatening bleeding.
Time Frame: Post-operative days 1, 3, and 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 15 | 24
score on a scale
  Post-operative day 1 | 1.5 (1.0) | 0.9 (0.6)
  Post-operative day 3 | 1.5 (1.0) | 0.9 (0.6)
  Post-operative day 7 | 0.7 (0.6) | 0.3 (0.5)

7. Post Hoc Outcome: Number of Mustache Gauze Changes
Description: Number of changes to post-operative wound dressing.
  This outcome was not collected based on difficulty with patient compliance. No data was gathered on this outcome measure.
Time Frame: Post operative days 1, 3 & 7
Population: No participants were analyzed
Arm/Group | Control | Ibuprofen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study period, which included the 7 days following sinus surgery.
Description: They do not differ from the clinical trials.gov definitions.
Arm/Group | Control | Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/26
Other Adverse Events (participants affected / at risk) | 0/16 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03055507/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT03055507/ICF_001.pdf